CLINICAL TRIAL: NCT02115269
Title: IndoProCaf (Difmetre®) Effervescent Tablets Effectiveness in Acute Treatment of Primary Headaches (Migraine and/or Episodic Tension-type Headache) and Patients' Satisfaction With the Treatment in Routine Clinical Practice in Ukraine and Kazakhstan
Brief Title: IndoProCaf Effervescent Tablets Effectiveness in Acute Treatment of Migraine and/or Episodic Tension-type Headache and Patients' Satisfaction With the Treatment in Routine Clinical Practice
Acronym: PRESTO
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Almedis (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-389
Record Dates: First submitted 2014-04-09; First posted 2014-04-16 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Headache Disorders, Primary; Migraine With Aura; Migraine Without Aura; Tension-Type Headache
Keywords: Indoprocaf; Indomethacin; Caffeine; Prochlorperazine; Migraine with Aura; Migraine without Aura; Tension-Type Headache
MeSH Terms: conditions — Headache Disorders, Primary; Migraine with Aura; Migraine without Aura; Tension-Type Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- primary headaches: Adults taking IndoProCaf for acute treatment of their primary headache attacks (migraine and/or episodic tension-type headache) as per routine clinical practice

SUMMARY:
Headaches are a common medical problem that physicians frequently encounter in their practice. One of key findings of The Atlas of Headache Disorders prepared by World Health Organization (WHO) is: headache disorders, including migraine and tension-type headache (TTH), are among the most prevalent disorders of mankind. The fixed combination of indomethacin, prochlorperazine and caffeine (IndoProCaf) showed efficacy and safety in acute treatment of migraine and episodic tension-type headache attacks. IndoProCaf (Difmetre®) is widely used in common daily practice only in Italy from early 1970s, is available at the Commonwealth of Independent States (CIS) pharmaceutical market now. There are limited data regarding IndoProCaf usage from post-marketing settings. This will be a first post-marketing observational study which aimed to evaluate the effectiveness and patients' satisfaction of primary headaches acute treatment in routine clinical settings in Ukraine and Kazakhstan.

DETAILED DESCRIPTION:
The study is designed as a prospective, multicentre, observational, non-interventional, non-randomized, non-controlled, single arm, post-marketing study where IndoProCaf will be prescribed in the usual manner per standard clinical practice of the treating physician and in accordance with the terms of the locally approved instruction for medical use. No additional procedures (other than the standard of care) shall be applied to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary headache (migraine with or without aura and/or episodic TTH) and whose headache attacks required acute pharmacological treatment.
* Were administered IndoProCaf (Difmetre®) effervescent tablets therapy according to the local product labelling.
* Adults 18 years and older (male, female).
* Provide Authorization to the investigator to use and/or disclose personal and/or health data.

Exclusion Criteria:

* Meet contraindications for treatment with IndoProCaf (Difmetre®) effervescent tablets as outlined in the latest version of local product labelling.
* Patients who are required prescription by physician of IndoProCaf and nonsteroidal anti-inflammatory drug-containing products at the same time for acute headache attacks treatment.
* Previous discontinuation of IndoProCaf treatment due to safety (i.e. hypersensitivity) events, lack of efficacy.
* Female patients who are pregnant or are breast-feeding.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with migraine (with or without aura) and/or episodic TTH
Sampling Method: Non-Probability Sample
Enrollment: 759 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Berrou, MD, Study Director — Abbott
Locations (30):
- Kazakhstan (15):
  - Research facility ID ORG-000986, Aktobe
  - LLP Medical Centre "Medical Assistance Group", Almaty
  - Research facility ID ORG-000994, Almaty
  - Research facility ID ORG-000990, Astana
  - Research facility ID ORG-000991, Astana
  - Research facility ID ORG-000992, Astana
  - State enterprise on the right of business City Clinic №1, Astana
  - LLP "State Center for Primary Health Care", Karaganda
  - LLP Clinic "Alanda", Karaganda
  - State enterprise on the right of business City Clinic №2, Karaganda
  - Branch of the JSC " Railway Hospital of the medical catastrophes" "Kostanay railway hospital", Kostanay
  - LLP "Aksim-plus", Kostanay
  - State enterprise on the right of business "Consultative-diagnostic center Semey", Semey
  - Research facility ID ORG-000989, Shymkent
  - State communal enterprise " City emergency health care hospital", Shymkent
- Ukraine (15):
  - Research facility ORG-001131, Dnipropetrovsk
  - Research facility ORG-001127, Kharkiv
  - Research facility ID ORG-000999, Kharkiv
  - Research facility ID ORG-000335, Kiev
  - "Public Institution ""Kyiv City Clinical Hospital №4"", Neurology Department №1 and №2;, Kyiv
  - "Public Institution 'Volyn Regional Clinical Hospital',, Lutsk
  - Research facility ID ORG-001001, Lviv
  - Research facility ID ORG-001004, Lviv
  - Research facility ID ORG-001000, Mukachevo
  - Research facility ID ORG-000340, Mykolaiv
  - Research facility ORG-001130, Odesa
  - Research faciity ID ORG-001003, Odesa
  - Research facility ORG-001129, Poltava
  - Education and Research Medical Center "University Hospital of Zaporizhzhia State Medical University", Neurology Department, Zaporizhzhia
  - Public Institution "Zaporizhzhia City Multispecialty Clinical Hospital №9", Neurology Department, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Headaches
Started | 759
Completed | 702
Not Completed | 57
Not completed — Lost to Follow-up | 43
Not completed — Did not complete patient diary | 3
Not completed — Moved to another city | 7
Not completed — Withdrawal by Subject | 2
Not completed — Didn't take study drug | 2

BASELINE CHARACTERISTICS:
Population: Safety set included all enrolled patients who have taken at least one dose of IndoProCaf
Arm/Group | Primary Headaches
Number analyzed (Participants) | 702
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 542
  Male | 160
Region of Enrollment [Count of Participants; unit: Participants]
  Ukraine | 432
  Kazakhstan | 270

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Significant Pain Reduction
Description: significant pain reduction defined as improvement to mild or no pain 2 hours post-dose by 4-point pain severity scale: 0 = no pain; 1 = mild headache, allowing normal activities; 2 = moderate headache, disturbing normal activities; 3 = severe headache, disabling activities, requiring bed-rest
Time Frame: up to 2 hours
Population: Number of patients in full analysis set. Full analysis set included all patients who signed informed consent and complied with all the inclusion and exclusion criteria and who had at least one acceptable headache attack treated with IndoProCaf documented in the patient's diary. This population was used for the effectiveness endpoints reporting.
Measure: Number; unit: percentage of participants
Arm/Group | Primary Headaches
Number analyzed (Participants) | 663
percentage of participants | 90.3

2. Primary Outcome: Percentage of Patients Who Are Satisfied With IndoProCaf Treatment
Description: Patients are asked to evaluate their satisfaction with headache pain reduction after treatment by selecting the options: =very poor, =poor, =no opinion, =good, =very good. The satisfied patients are defined as those with =good and = very good answers.
Time Frame: up to 24 hours post dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Primary Headaches
Number analyzed (Participants) | 663
percentage of participants | 91.3

3. Secondary Outcome: Time to Significant Pain Reduction
Description: Time to significant pain reduction at 1, 2, 4, 6 and 24 hours post-dose period are summarized with number of patients in each category; significant pain reduction is defined as improvement to mild or no pain 2 hours post-dose by 4-point pain severity scale: 0 = no pain; 1 = mild headache, allowing normal activities; 2 = moderate headache, disturbing normal activities; 3 = severe headache, disabling activities, requiring bed-rest
Time Frame: up to 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Significant Pain Reduction at 1 Hour Post Dose: Adults taking IndoProCaf for acute treatment of their primary headache attacks (migraine and/or episodic tension-type headache) as per routine clinical practice and achieved significant pain reduction at 1 hour post dose
- Significant Pain Reduction at 2 Hours Post Dose: Adults taking IndoProCaf for acute treatment of their primary headache attacks (migraine and/or episodic tension-type headache) as per routine clinical practice and achieved significant pain reduction at 2 hours post dose
- Significant Pain Reduction at 4 Hour Post Dose: Adults taking IndoProCaf for acute treatment of their primary headache attacks (migraine and/or episodic tension-type headache) as per routine clinical practice and achieved significant pain reduction at 4 hours post dose
- Significant Pain Reduction at 6 Hours Post Dose: Adults taking IndoProCaf for acute treatment of their primary headache attacks (migraine and/or episodic tension-type headache) as per routine clinical practice and achieved significant pain reduction at 6 hours post dose
- Significant Pain Reduction at 24 Hours Post Dose: Adults taking IndoProCaf for acute treatment of their primary headache attacks (migraine and/or episodic tension-type headache) as per routine clinical practice and achieved significant pain reduction at 24 hours post dose
Arm/Group | Significant Pain Reduction at 1 Hour Post Dose | Significant Pain Reduction at 2 Hours Post Dose | Significant Pain Reduction at 4 Hour Post Dose | Significant Pain Reduction at 6 Hours Post Dose | Significant Pain Reduction at 24 Hours Post Dose
Number analyzed (Participants) | 663 | 663 | 663 | 663 | 663
participants | 464 | 252 | 176 | 50 | 15

4. Secondary Outcome: Percentage of Patients With Significant Pain Reduction in Case of First Dose no Response
Description: as for outcome 1
Time Frame: up to 2 hours
Population: Patients who took second IndoProCaf dose at 2 hours post-dose
Measure: Number; unit: percentage of participants
Arm/Group | Primary Headaches
Number analyzed (Participants) | 225
percentage of participants | 55.6

5. Secondary Outcome: Percentage of Patients With Significant Pain Reduction in Case of Headache Relapse
Description: as for outcome 1
Time Frame: up to 48 hours
Population: Patients who had headache relapse. Headache relapse was defined as a worsening of headache attack after 24 hours of the initial dosing and pain-free at 2h but no later than 48 hours of initial IndoProCaf dosing.
Measure: Number; unit: percentage of participants
Arm/Group | Primary Headaches
Number analyzed (Participants) | 80
percentage of participants | 90.0

6. Secondary Outcome: Percentage of Patients Who Are Satisfied With Different Medicines Previously Used for Headache Attack
Description: Defined as good and very good by Likert-type scale (e.g. very poor, poor, no opinion, good, very good)
Time Frame: baseline
Population: Patients who took trip tans in the past (data are from Safety set which included all enrolled patients who have taken at least one dose of IndoProCaf).
Measure: Number; unit: percentage of participants
Groups:
- Patients With Primary Headaches and Took Triptans in the Past: Adults taking IndoProCaf for acute treatment of their primary headache attacks (migraine and/or episodic tension-type headache) as per routine clinical practice who took triptans in the past.
- Patients With Primary Headaches Who Took NSAIDs and Analgesics: Adults taking IndoProCaf for acute treatment of their primary headache attacks (migraine and/or episodic tension-type headache) as per routine clinical practice and who took NSAIDs and analgesics
- Patients Who Took Combined Analgesics: Adults taking IndoProCaf for acute treatment of their primary headache attacks (migraine and/or episodic tension-type headache) as per routine clinical practice and who took combined analgesics in the past
- Patients Who Took Ergotamine-based Drugs: Adults taking IndoProCaf for acute treatment of their primary headache attacks (migraine and/or episodic tension-type headache) as per routine clinical practice and who took ergotamine-based drugs in the past
- Patients Who Took Antiemetics: Adults taking IndoProCaf for acute treatment of their primary headache attacks (migraine and/or episodic tension-type headache) as per routine clinical practice and who took antiemetics in the past
- Patients Who Took Opioid Analgesics: Adults taking IndoProCaf for acute treatment of their primary headache attacks (migraine and/or episodic tension-type headache) as per routine clinical practice and who took opioid analgesics in the past
Arm/Group | Patients With Primary Headaches and Took Triptans in the Past | Patients With Primary Headaches Who Took NSAIDs and Analgesics | Patients Who Took Combined Analgesics | Patients Who Took Ergotamine-based Drugs | Patients Who Took Antiemetics | Patients Who Took Opioid Analgesics
Number analyzed (Participants) | 128 | 515 | 387 | 34 | 34 | 11
percentage of participants | 48.4 | 22.1 | 29.2 | 35.3 | 23.5 | 27.3

ADVERSE EVENTS:
Description: Overall 33 Adverse Events (AEs) were reported in 19 (2.7%) patients who participated in this study. Three (3) events were serious. There were no AEs that exceeded 5% frequency threshold.
  The most frequent (AEs) by System Organ Class (SOC) were gastrointestinal disorders and nervous system disorders, 9 AEs in 7 (1%) patients were reported in each of these groups.
Arm/Group | Primary Headaches
Serious Adverse Events (participants affected / at risk) | 3/702
Other Adverse Events (participants affected / at risk) | 16/702
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Headaches (N=702)
Hypertension crisis (Vascular disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Loss of consiousness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Headaches (N=702)
Nausea (Gastrointestinal disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Visual impairment (Eye disorders) | 3 (3)
Asthenia (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Blood pressure increased (Investigations) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less